CLINICAL TRIAL: NCT01988272
Title: Imaging Based Dosimetry for Individualized Internal Emitter Therapy
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Yuni Dewaraja, Research Associate Professor, University of Michigan
Other Study IDs: 5R01EB001994 (NIH)
Record Dates: First submitted 2013-11-05; First posted 2013-11-20 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: SPECT/CT; Dosimetry; Radiation absorbed dose; Non-Hodgkin's Lymphoma; I-131 tositumomab radioimmunotherapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: SPECT/CT imaging — Patients will undergo scanning on the above system.
  Other Names: Siemens Symbia SPECT/CT system

SUMMARY:
The goal of this study is to develop imaging based methods to accurately determine the energy absorbed (absorbed dose) by tumor tissue and bone marrow after radioimmunotherapy with I-131 tositumomab . The administration of the radioactive, iodine-131 labeled, monoclonal antibody I-131 tositumomab, (also known as Bexxar) is part of the patient's clinical treatment protocol. For the absorbed dose measurement, investigators at the University of Michigan are evaluating a new Nuclear Medicine SPECT/CT imaging system . This new camera combines a CT imaging system in addition to a Nuclear Medicine SPECT scanner. CT scans allow the doctors to see a high quality picture of your internal organs. The Nuclear Medicine SPECT scanner allows the doctors to see the uptake of the radioactive I-131 including the tumor sites. The improved imaging using the SPECT/CT enables more accurate calculation of the energy absorbed by tumor tissue and bone marrow. Using the results from these calculations and clinical follow up data, the researchers will investigate the relationship between the absorbed dose to the tumor and the patient's tumor response as well as the relationship between the absorbed dose to the bone marrow and the bone marrow toxicity. These relationships can potentially be used in the future by doctors to help determine how much radioactive I-131 to administer to each patient to get optimal results.

ELIGIBILITY:
Inclusion Criteria:

* • Clinically stable patients undergoing I-131 Tositumomab (Bexxar) for treatment of Non-Hodgkin Lymphomas

Exclusion Criteria:

* • Clinical instability

  * Patients who are unable to lie flat on the imaging systems long enough to permit imaging protocols to be performed
  * Refusal to provide informed consent
  * Patients who are pregnant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically stable patients undergoing I-131 Tositumomab (Bexxar) for treatment of Non-Hodgkin Lymphomas
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-06; Primary Completion 2015-03 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Correlation between radiation absorbed dose to tumor and response or progression free survival | 6 months
  Tumor absorbed doses will be calculated based on research SPECT/CT imaging and correlated with the response as assessed by clinical PET/CT.

SECONDARY OUTCOMES:
Assess correlation between radiation absorbed dose to the bone marrow and hematologic toxicity. | 6 months
  Absorbed dose will be determined by SPECT/CT imaging of the marrow rich lumbar region and will be correlated with toxicity based on follow-up blood counts.

CONTACTS AND LOCATIONS:
Overall Officials: Yuni Dewaraja, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States